CLINICAL TRIAL: NCT05943938
Title: Prospective Evaluation of Sepsis Prediction Algorithms in a Multi-Hospital Healthcare System
Brief Title: Comparison of Sepsis Prediction Algorithms
Status: Not yet recruiting | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Siva Bhavani, Assistant Professor, Emory University
Other Study IDs: STUDY00005958; 2024P008316 (Other: Emory IRB)
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Sepsis
Keywords: Infection; Emergency Department; Algorithm; Prediction
MeSH Terms: conditions — Sepsis; Infections; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ED Patients: All adult patients presenting to Emergency Departments (ED) in the Emory Healthcare system
  Interventions: Other: Epic Sepsis Model Version - 1; Other: Epic Sepsis Model Version - 2; Other: Emory Sepsis Model

INTERVENTIONS:
Other: Epic Sepsis Model Version - 1 — The Epic Sepsis Model (ESM) version 1, a proprietary sepsis prediction model.
  Other Names: Proprietary Epic sepsis algorithm -1
Other: Epic Sepsis Model Version - 2 — The Epic Sepsis Model (ESM) version 2, a proprietary sepsis prediction model.
  Other Names: Proprietary Epic sepsis algorithm -2
Other: Emory Sepsis Model — Emory internal algorithm
  Other Names: Emory Sepsis Algorithm

SUMMARY:
Sepsis is a severe response to infection resulting in organ dysfunction and often leading to death. More than 1.5 million people get sepsis every year in the U.S., and 270,000 Americans die from sepsis annually. Delays in the diagnosis of sepsis lead to increased mortality. Several clinical decision support algorithms exist for the early identification of sepsis. The research team will compare the performance of three sepsis prediction algorithms to identify the algorithm that is most accurate and clinically actionable. The algorithms will run in the background of the electronic health record (EHR) and the predictions will not be revealed to patients or clinical staff. In this current evaluation study, the algorithms will not affect any part of a patient's care. The algorithms will be deployed across the Emory healthcare system on data from all patients presenting to the emergency department.

DETAILED DESCRIPTION:
The primary goal of this study is to prospectively evaluate three sepsis prediction algorithms that are embedded in the EHR. The models will be deployed in a "shadow" mode, and the results will not be displayed to the treatment team during this study. Two of the algorithms are proprietary algorithms of the EHR provider (Epic). The third algorithm is an internally developed, open-source algorithm.

The algorithms will compute the probability of sepsis at periodic intervals and will continue to run on a patient's data until the patient's discharge, death, or upon initiation of intravenous antibiotics (at which point there is an indirect record of clinical suspicion of an infection).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted through the ED

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted through the ED from the time they arrive at the hospital until discharge, death, or initiation of intravenous antibiotics.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient hospitalization-level area under curve (AUC) for identification of sepsis, | Duration of hospital stay (until discharge or death), an expected average of 30 days
  Definition of Sepsis using the Centers for Disease Control and Prevention (CDC) Adult Sepsis Surveillance.

SECONDARY OUTCOMES:
Sensitivity, specificity, and Positive and Negative Predictive Value of algorithms | Duration of hospital stay (until discharge or death), an expected average of 30 days
  Sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV).
Lead time to antibiotic administration | Duration of hospital stay (until discharge or death), an expected average of 30 days
  The time between the initial deployment of the alert in patients confirmed to have sepsis (ture positives) and the physician's ordering of intravenous antibiotic therapy.
Percent expected increase in unnecessary antibiotics | Duration of hospital stay (until discharge or death), an expected average of 30 days
  Percent of patients who were incorrectly identified as having sepsis (false positives), and received antibiotics.
Number needed to screen | Duration of hospital stay (or death), an expected average of 30 days
  The number of alerts that would need to be processed to find one true positive sepsis.
Number of Total and false alert burden | Duration of hospital stay (until discharge or death), an expected average of 30 days
  The number of Total and false alert burden cumulative across all study patients over the study period
Time-horizon based AUCs | 4 hours, 8 hours, and 24 hours
  AUCs will be calculated at 3 pre-specified time horizons.
Accuracy and calibration by subgroup | Duration of hospital stay (until discharge or death), an expected average of 30 days
  The AUC and calibration curves will be compared by sex and race to ensure predictive accuracy is equal across subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Sivasubramanium Bhavani, MD, Principal Investigator — Emory University
Locations (7):
- United States (7):
  - Emory Midtown Hospital, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Healthcare System, Atlanta, Georgia
  - Emory Hospital, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Emory Hillandale Hospital, Lithonia, Georgia

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share individual participant data that underlie the results reported in an article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Data will be shared beginning 6 months after publication, without a specified end date.
Access Criteria: To gain access, data requestors will need to sign a data access agreement.